CLINICAL TRIAL: NCT05014009
Title: The Influence of Neuromuscular Training on Whole-body Movement Strategies and Knee Mechanics During Change-of-direction Tasks in Sports Science Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: University of Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Maurice Mohr, Principal Investigator, Universitaet Innsbruck
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2107COD
Record Dates: First submitted 2021-08-06; First posted 2021-08-20 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: electromyography; inertial measurement unit; neuromuscular training; muscle activity; muscle synergy; sidestepping movement; side-cutting movement
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to multidirectional training group (MD) or a linear sprint training group (LS) in a quasi-randomized way. Both groups will complete an 8-week training program and will complete baseline, follow-up, and retention testing (4 weeks post follow-up).
Masking Description: While the study team will not point participants to the specific differences between the two training programs (MD vs. LS), an exchange between participants about the training elements in each group cannot be avoided given that the participants are all students at the same faculty. Given that the study team will supervise the training sessions, collect the data, and assess the outcomes, blinding of investigators will not be possible but the analysis will be designed to minimize sources of investigator bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA11+ and multidirectional training (MD) (Experimental): Participants in the MD group will take part in an 8-week NMT intervention known to reduce the risk of sports injury and expected to improve COD movement strategies.
  Interventions: Behavioral: FIFA11+ and multidirectional training (MD)
- FIFA11+ and linear sprint training (LS) (Active Comparator): Participants in the LS group will take part in an 8-week NMT intervention, which is known to reduce the risk of sports injury but is unlikely to improve COD movement strategies and is expected to improve linear sprint performance.
  Interventions: Behavioral: FIFA11+ and linear sprint training (MD)

INTERVENTIONS:
Behavioral: FIFA11+ and multidirectional training (MD) — This intervention initially contains a shortened version of the FIFA11+ injury prevention program including running (straight, hip out, hip in, jump-run-ups), strengthening (planks, squats, nordic hamstring curls), and single-leg balance exercises. The initial part is followed by COD technique modification training, which contains exercises aimed at improving COD technique (safer and more effective body re-direction, use of penultimate step, avoiding knee valgus) and COD braking and re-acceleration impulse.
  The duration of each training session is 25-30 minutes. The training is carried out twice per week under supervision with supervisors providing feedback to participants regarding their COD technique. Participants are encouraged to complete a third training session in their own time.
  Arms: FIFA11+ and multidirectional training (MD)
Behavioral: FIFA11+ and linear sprint training (MD) — This intervention initially contains a shortened version of the FIFA11+ injury prevention program including running (straight, hip out, hip in, jump-run-ups), strengthening (planks, squats, nordic hamstring curls), and single-leg balance exercises. The initial part is followed by a linear sprint training, which contains exercises aimed at improving sprint technique (e.g. sagittal arm and leg movement, trunk lean), use of the stretch-shortening cycle, leg stiffness and propulsive impulse .
  The duration of each training session is 25-30 minutes. The training is carried out twice per week under supervision with supervisors providing feedback to participants regarding their sprinting technique. Participants are encouraged to complete a third training session in their own time.
  Arms: FIFA11+ and linear sprint training (LS)

SUMMARY:
Background

Knee injuries are common during sports that require fast change-of-direction (COD) movements such as sidestepping and pivoting during soccer, basketball, handball, and related sports. COD movements expose the knee joint to large external forces, particularly if players show a poor COD technique such as lateral trunk lean towards the plant foot or a strong knee valgus of the cutting leg. Larger external forces and moments that act on the knee joint are expected to result in larger strain of the anterior cruciate ligament (ACL) and thus a higher risk of ACL rupture. Consequently, during sports like soccer and basketball, many non-contact ACL injuries occur during COD tasks. While neuromuscular training (NMT) programs have been developed to effectively reduce the risk of sports injury including ACL tears, ACL injury rates have not declined in the last years. One of the reasons for this paradox may be that many NMT programs such as the FIFA11+ program, which were developed to protect from injury do not actually improve COD movement strategies. It may be assumed that FIFA11+ does reduce the overall risk of sports injury through general improvements in strength and balance as well as safer jump landing technique but not through safer COD technique. Further, if training interventions were successful in reducing 'high-risk' movement patterns and in developing knee-stabilizing muscle synergies during COD movements, it remains unclear whether the improved movement strategy, e.g. the reduction in external knee valgus moments, actually corresponds to reduced ACL strain. In consequence, there is the need for a comprehensive investigation to determine whether a NMT program focused on improving COD technique will improve COD movement and muscle activation strategies and whether these improvements are correlated with estimated ACL strain.

A second reason for the paradox may be that current experimental protocols to investigate COD movement strategies in the laboratory are not a good indicator for actual player behavior on the field thus masking potential benefits of NMT on lateral movements. Therefore, the sports injury prevention community should aim to move the assessment of COD movement strategy onto the playing field and into a more realistic playing environment while characterizing the kinematics and kinetics of sidestepping based on wearable sensors. In consequence, novel analytical frameworks based on wearables need to be developed, which can capture full-body kinematics and the underlying forces during COD movements on the playing field. In the long run, such systems could facilitate real-time feedback with respect to COD technique on the playing field and thus enhance motor learning of the players as well as characterize real-world player agility.

Research objectives & hypotheses

Objective 1: To determine the effect of an 8-week NMT and COD technique modification intervention (multidirection training, MD) on 1) COD movement strategies as characterized by the lateral trunk angle and knee valgus moment and 2) estimated ACL strain during 45- and 135-degree COD movements in comparison to an 8-week NMT and linear sprint training intervention (linear sprint training, LS) in sports science students.

Hypothesis 1: There will be a larger reduction in lateral trunk angle and knee valgus moment and an associated reduction in ACL strain in the MD group compared to the LS group following the 8-week intervention, which will be retained four weeks later.

Objective 2: To determine the effect of an 8-week NMT and COD technique modification intervention on leg muscle synergies as characterized by the number of muscles and the structure of the synergy vector for each identified muscle synergy in comparison to an 8-week NMT and linear sprint training intervention in sports science students.

Hypothesis 2: One or multiple muscle synergy vectors will show an increased contribution of hip abductor muscle activity in the MD group following training and there will be a lower number of activated muscles per identified synergy, i.e. a more selective muscle activation in comparison to the LS group. These improvements will be retained four weeks later.

Objective 3: To determine the validity of an analysis framework to estimate COD movement strategy (lateral trunk angle, foot progression angle, knee valgus moment) and ACL strain based solely on inertial motion capture data in comparison to the gold-standard of 3D optimal motion capture.

DETAILED DESCRIPTION:
Study design and participants

This is a quasi-randomized trial to investigate the effects of effects of two neuromuscular training interventions (multidirectional vs. linear sprint training) on COD movement strategies in sports science students and in parallel to develop a methodological framework for field-based COD movement assessments. This trial will be registered with ClinicalTrials.gov after ethical approval has been granted. An a-priori sample size estimation was conducted based on a previous non-randomized controlled trial reporting a strong, beneficial effect of a 6-week COD technique modification on the Cutting Movement Assessment Score (CMAS), a qualitative screening tool to quantify biomechanical and neuromuscular deficits during COD tasks [significant group x time interaction, Cohen's f2 = 0.63 (right leg) - 1.00 (left leg)]. With an a-priori significance level of alpha = 0.05 and a desired power of 0.8, the minimum required sample size was estimated in G*Power v3.1.9.7 as only N = 8 (n = 4 in each training group). One concern with this previous study is, however, that CMAS raters were not blinded to group assignment leading to a potential systematic bias and overestimated effect size. A second concern is that the CMAS, which combines multiple biomechanical and neuromuscular deficits (e.g. knee valgus, lateral trunk flexion, hip internal rotation) into one aggregate score may show a larger effect compared to the analysis of single biomechanical variables (e.g. knee abduction moment) like in the current study. Based on these considerations the required sample size of N = 40 sports science students (n = 20 for the MD and LS) was selected. With an expected drop-out rate of 25%, this sample of at least N = 30 participants will enable to detect moderate to strong interaction effects (Cohen's f2 > 0.3) with a power of at least 0.8.

Experimental protocol

All participants will take part in a first familiarization session (WN 40) to practice the execution of the COD task and receive information about the content and goals of the training intervention. Baseline testing (WN 40-41), follow-up testing (WN 49-50), and retention testing (WN2-4, 2022) will be conducted in the laboratory Pulverturm at the ISW Innsbruck and will follow the same testing protocol. Participants will be equipped with 47 retroreflective markers for 3D motion analysis (extended full-body PlugIn Gait model, 10 cameras, 200 Hz) and 14 sensors for combined measurements of surface electromyography (sEMG, 2000 Hz) and inertial segment data (200 Hz) (Noraxon Ultium, Noraxon Inc., Scottsdale, AZ, USA) of the right leg. Afterwards, the participants will be asked to warm-up on a stationary bike for five minutes followed by the initial running exercises of the FIFA11+ program. Maximum voluntary contractions (MVCs) will be obtained for ankle plantarflexion/dorsiflexion, knee flexion/extension, hip extension/flexion, and hip abduction according to standardized manual tests. IMU position and orientation with respect to the participants' anatomy will be determined based on images and calibration movements taken before the start of the measurements. After four successful practice trials, participants will be asked to complete 10 COD movements with a 45-degree cutting angle (COD45) and 10 COD movements with a 135-degree cutting angle (COD135) always planting and cutting with the right foot on a ground-embedded force plate (1000 Hz, Kistler, Winterthur, Switzerland). The approach and exit speed for each COD movement will be controlled to approximately 4.5 m/s (COD45) and 4 m/s (COD135) as measured by optical timing gates placed within the approach and exit zones (Witty, Microgate, Bolzano, Italy). Rest periods of one minute in between trials and five minutes in between blocks (COD45 vs. COD135) will avoid accumulation of neuromuscular fatigue.

Data analysis

Using the 3D marker trajectories and force data as inputs (optimal motion capture, OMC, model), full-body kinematics, 3D joint moments, muscle forces, and ACL strain will be estimated using inverse kinematics and EMG-informed optimization procedures in OpenSim (v.4.2) combined with FE simulations.

Using only the inertial sensor data as inputs (inertial motion capture, IMC, model), full-body kinematics, 3D joint moments, muscle forces, and ACL strain will be estimated using an IMU-tracking and optimal control algorithm combined with FE simulations. This latter approach is novel and is currently being developed.

The muscle activation pattern of the right leg will be further analyzed via a muscle synergy analysis [one muscle synergy model for each testing time point (baseline, follow-up 1, follow-up 2] and quantified according to its muscle synergy vectors and synergy activation profiles. Specifically, the number of muscles per synergy vector and the shape of the muscle synergy vectors will serve as additional dependent variables.

Statistics

Objective 1 & 2: Effects of the NMT and COD technique modification intervention on the kinematic, kinetic (OMC model), and EMG-related outcome variables will be tested according to a repeated measures ANOVA with the between-subject factor 'group' (MD vs. LS) and the within-subject factor 'time point' (baseline, follow-up, retention). The null hypothesis H1 will be rejected if there is a significant interaction effect 'group x time point' at an a-priori significance level of alpha = 0.05. Interaction effects, i.e. effect modification, due to the participants' sex or potential other covariates (e.g. baseline COD performance) will be explored in additional three-way repeated measures ANOVAs. Post-hoc testing will investigate changes in dependent variables between time points for each group.

Objective 3: The validity of the IMC model will be determined based on Bland & Altman limits of agreement to estimate the systematic bias and random error of the IMC model-based dependent variables in comparison to the OMC model-based variables. The IMC model will be called valid if the limits of agreement are smaller than the observed changes in the corresponding variables between baseline and follow-up testing in the intervention group.

Ethical considerations / risk-benefit analysis / insurance information

All participants will be sports science students and thus frequently encounter the injury risks associated with multi-directional sports. Therefore, the risk of injury for participants in this study will be no higher than in their everyday life. In the rare case that a participant sustains an injury during this study, he/she will be covered by accident insurance provided to all University of Innsbruck students. Furthermore, all participants will benefit from participating in the current study given that the FIFA11+ NMT program, which is part of the training in both training groups, has been shown to effectively reduce the risk of sports injury. Overall, the benefits of this study outweigh the risks.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a student at the Department of Sport Science in Innsbruck

Exclusion Criteria:

* Clinical diagnosis of a lower extremity muscle or joint injury within the last six months that led to a disruption of sport participant by at least two weeks
* Clinical diagnosis of a balance disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Peak knee abduction moment in Nm assessed through 3D optical motion capture | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  Peak external knee moment in the frontal plane during the COD stance phase
Peak lateral trunk lean in degrees assessed through 3D optical motion capture | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  Peak angle of the trunk with respect to a vertical line in the frontal plane during the COD stance phase. Of interest is the angle opposite to the direction of intended travel.
Peak ACL strain in % estimated through finite element simulation | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  Peak ACL strain estimated from the EMG-informed musculoskeletal and FE simulation.

SECONDARY OUTCOMES:
Muscle synergy size (number of muscles per synergy) assessed through non-negative matrix factorization of the surface EMG data | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  The average number of muscles across identified muscle synergies during the COD stance phase.
Hip muscle contribution in % assessed through non-negative matrix factorization of the surface EMG data | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  The synergy vector coefficients of the hip muscles (rectus femoris, semitendinosus, biceps femoris, gluteus medius) within each identified muscle synergy
Linear sprint performance in seconds assessed through a timing gate system | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  Time in a 10m standing start sprint
COD performance in seconds assessed through a timing gate system | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  Time to complete a 45 deg and 135 deg change-of-direction drill

OTHER OUTCOMES:
Peak knee abduction moment in Nm assessed through inertial motion capture | Assessed in October (baseline), December (follow-up), February (retention) over a total duration of 5 months.
  Peak external knee moment in the frontal plane during the COD stance phase from the IMU-based analysis approach

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Mohr, PhD, Principal Investigator — University of Innsbruck, Austria
Locations (1):
- Department of Sport Science, University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Yes
The raw data (motion capture, EMG, and anonymous participant information) will be shared via an open access data repository along with the publications that present the study results.
Time Frame: Data will be shared via an open access data repository along with the publications that present the study results.
Access Criteria: Open access

REFERENCES:
- [Background] Turpin NA, Uriac S, Dalleau G. How to improve the muscle synergy analysis methodology? Eur J Appl Physiol. 2021 Apr;121(4):1009-1025. doi: 10.1007/s00421-021-04604-9. Epub 2021 Jan 26. PMID 33496848
- [Background] McLean SG, Huang X, Su A, Van Den Bogert AJ. Sagittal plane biomechanics cannot injure the ACL during sidestep cutting. Clin Biomech (Bristol). 2004 Oct;19(8):828-38. doi: 10.1016/j.clinbiomech.2004.06.006. PMID 15342155
- [Background] Benjaminse A, Gokeler A, Dowling AV, Faigenbaum A, Ford KR, Hewett TE, Onate JA, Otten B, Myer GD. Optimization of the anterior cruciate ligament injury prevention paradigm: novel feedback techniques to enhance motor learning and reduce injury risk. J Orthop Sports Phys Ther. 2015 Mar;45(3):170-82. doi: 10.2519/jospt.2015.4986. Epub 2015 Jan 27. PMID 25627151
- [Background] Delp SL, Anderson FC, Arnold AS, Loan P, Habib A, John CT, Guendelman E, Thelen DG. OpenSim: open-source software to create and analyze dynamic simulations of movement. IEEE Trans Biomed Eng. 2007 Nov;54(11):1940-50. doi: 10.1109/TBME.2007.901024. PMID 18018689
- [Background] Dempsey AR, Lloyd DG, Elliott BC, Steele JR, Munro BJ. Changing sidestep cutting technique reduces knee valgus loading. Am J Sports Med. 2009 Nov;37(11):2194-200. doi: 10.1177/0363546509334373. Epub 2009 Jun 9. PMID 19509415
- [Background] Donnelly CJ, Lloyd DG, Elliott BC, Reinbolt JA. Optimizing whole-body kinematics to minimize valgus knee loading during sidestepping: implications for ACL injury risk. J Biomech. 2012 May 11;45(8):1491-7. doi: 10.1016/j.jbiomech.2012.02.010. Epub 2012 Mar 3. PMID 22387123
- [Background] Dorschky E, Nitschke M, Seifer AK, van den Bogert AJ, Eskofier BM. Estimation of gait kinematics and kinetics from inertial sensor data using optimal control of musculoskeletal models. J Biomech. 2019 Oct 11;95:109278. doi: 10.1016/j.jbiomech.2019.07.022. Epub 2019 Aug 1. PMID 31472970
- [Background] Dos'Santos T, McBurnie A, Comfort P, Jones PA. The Effects of Six-Weeks Change of Direction Speed and Technique Modification Training on Cutting Performance and Movement Quality in Male Youth Soccer Players. Sports (Basel). 2019 Sep 6;7(9):205. doi: 10.3390/sports7090205. PMID 31489929
- [Background] Emery CA, Roy TO, Whittaker JL, Nettel-Aguirre A, van Mechelen W. Neuromuscular training injury prevention strategies in youth sport: a systematic review and meta-analysis. Br J Sports Med. 2015 Jul;49(13):865-70. doi: 10.1136/bjsports-2015-094639. PMID 26084526
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Krosshaug T, Nakamae A, Boden BP, Engebretsen L, Smith G, Slauterbeck JR, Hewett TE, Bahr R. Mechanisms of anterior cruciate ligament injury in basketball: video analysis of 39 cases. Am J Sports Med. 2007 Mar;35(3):359-67. doi: 10.1177/0363546506293899. Epub 2006 Nov 7. PMID 17092928
- [Background] Lockie RG, Murphy AJ, Callaghan SJ, Jeffriess MD. Effects of sprint and plyometrics training on field sport acceleration technique. J Strength Cond Res. 2014 Jul;28(7):1790-801. doi: 10.1519/JSC.0000000000000297. PMID 24149762
- [Background] Markolf KL, Burchfield DM, Shapiro MM, Shepard MF, Finerman GA, Slauterbeck JL. Combined knee loading states that generate high anterior cruciate ligament forces. J Orthop Res. 1995 Nov;13(6):930-5. doi: 10.1002/jor.1100130618. PMID 8544031
- [Background] Oliveira AS, Silva PB, Lund ME, Farina D, Kersting UG. Balance Training Enhances Motor Coordination During a Perturbed Sidestep Cutting Task. J Orthop Sports Phys Ther. 2017 Nov;47(11):853-862. doi: 10.2519/jospt.2017.6980. Epub 2017 Sep 23. PMID 28944715
- [Background] Rajagopal A, Dembia CL, DeMers MS, Delp DD, Hicks JL, Delp SL. Full-Body Musculoskeletal Model for Muscle-Driven Simulation of Human Gait. IEEE Trans Biomed Eng. 2016 Oct;63(10):2068-79. doi: 10.1109/TBME.2016.2586891. Epub 2016 Jul 7. PMID 27392337
- [Background] Thompson JA, Tran AA, Gatewood CT, Shultz R, Silder A, Delp SL, Dragoo JL. Biomechanical Effects of an Injury Prevention Program in Preadolescent Female Soccer Athletes. Am J Sports Med. 2017 Feb;45(2):294-301. doi: 10.1177/0363546516669326. Epub 2016 Oct 29. PMID 27793803
- [Background] Ueno R, Navacchia A, Schilaty ND, Myer GD, Hewett TE, Bates NA. Anterior Cruciate Ligament Loading Increases With Pivot-Shift Mechanism During Asymmetrical Drop Vertical Jump in Female Athletes. Orthop J Sports Med. 2021 Mar 9;9(3):2325967121989095. doi: 10.1177/2325967121989095. eCollection 2021 Mar. PMID 34235227
- [Background] Walden M, Hagglund M, Magnusson H, Ekstrand J. ACL injuries in men's professional football: a 15-year prospective study on time trends and return-to-play rates reveals only 65% of players still play at the top level 3 years after ACL rupture. Br J Sports Med. 2016 Jun;50(12):744-50. doi: 10.1136/bjsports-2015-095952. Epub 2016 Mar 31. PMID 27034129
- [Background] Young W, Rayner R, Talpey S. It's Time to Change Direction on Agility Research: a Call to Action. Sports Med Open. 2021 Feb 12;7(1):12. doi: 10.1186/s40798-021-00304-y. PMID 33580424
- See also: FIFA11+ Manual [in GERMAN] — https://www.dfb.de/fileadmin/_dfbdam/16988-Elf-Plus-Manual-Deutsch.pdf